CLINICAL TRIAL: NCT07032155
Title: The Feasibility of Implementing Virtual Reality-based Upper Limb Rehabilitation for Stroke Patients and Occupational Therapists in an Acute Stroke Unit and Community Stroke Team, in Terms of Technology Acceptance, Safety and Usability
Brief Title: Virtual Reality in Occupational Therapy Upper Limb Stroke Rehabilitation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: eXRt Intelligent Healthcare (Industry)
Collaborators: Belfast Health and Social Care Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EIHCT001
Record Dates: First submitted 2025-06-05; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stroke survivor participant group (Active Comparator): Participants receive VR therapy 30mins of the intervention 3 times a week for 4 weeks
  Interventions: Device: Resynk VR session
- Occupational therapist Participant group (Other): Occupational therapist Participants receive training and use VR on stroke survivor participants
  Interventions: Other: Using Resynk VR on stroke survivors

INTERVENTIONS:
Device: Resynk VR session — The study will use hardware and software to achieve this immersive virtual reality. The Resynk Virtual Reality programme (software) and the Meta Quest Virtual Reality Headset (hardware) will be used. Immersive virtual reality (VR) is when technology makes you feel like you're inside a different world. You wear a virtual reality headset that covers your eyes and ears, showing you a 3D world and playing matching sounds. The headset's head tracking, changing the view in the VR world as you look around. You can then interact with this virtual reality world depending on the application or game you use. The Resynk VR software launches automatically, guiding them through therapist-designed games that make rehabilitation engaging. The system uses advanced hand-tracking technology, eliminating the need for physical controllers. It detects joint movements in the hands and fingers, allowing users to perform key rehabilitation exercises such as supination, pronation, grasping, and pinching.
  Arms: stroke survivor participant group
Other: Using Resynk VR on stroke survivors — The Resynk Virtual Reality programme (software) and the Meta Quest Virtual Reality Headset (hardware) will be used by Occupational therapy participants to treat the stroke survivor participants
  Arms: Occupational therapist Participant group

SUMMARY:
The study aims to assess the feasibility of using Resynk, a virtual reality (VR) software platform for upper limb rehabilitation for stroke survivors, both in acute hospital settings and in the community (home, private nursing home, residential home). Resynk offers interactive, task-oriented training that enhances therapy intensity and patient motivation. Previous findings from a Quality Improvement project showed significant increases in treatment intensity and patient engagement with Resynk. This study will explore barriers to Resynk implementation and gather input from staff participants and stroke survivors to ensure successful integration and effectiveness.

Resynk will be delivered alongside standard care, with no intention to delay or reduce existing rehabilitation services. The study involves two participant groups -adult stroke survivors and Occupational Therapists. These represent realistic and appropriate user groups for this stage of implementation research. A control group is not included, as the primary aim is not comparative effectiveness but to assess feasibility and user experience.

This study will use a exploratory approach to using qualitative methods for gather insight into safety, acceptability and usability such as the System usability Scale, EQ-5D-5L and custom design Questionnaire. Quantitative methods will be used for evaluating rehabilitating and function outcomes this includes data collected by the Resynk application and the standardised Fugl Meyers assessment. The study will involve pre, post and follow up data collection for both participant groups.

ELIGIBILITY:
Inclusion Criteria:

Stroke Participants

Able to provide informed consent

Aged over 18 years.

Evidence of stroke confirmed by medical team

Newly diagnosed patients who are admitted to the acute stroke unit with a confirmed diagnosis of stroke.

More than 48 hours since stroke event

Patient is appropriate to participate in rehabilitation according to the treating physician or medical consultant, and able to follow simple verbal commands.

Presence of an upper limb deficit identified in the NIHSS (National Institutes of Health Stroke Scale) or by a member of the medical or multidisciplinary team

Residents within the Belfast health and social care trust catchment area/postcode

Staff participants:

Qualified Registered Occupational Therapy Staff who work in the Stroke Unit in the Royal Victoria Hospital Belfast or in the Community Stroke Team in the Belfast Health and Social Care Trust.

Able to provide informed consent

Aged 18 or over

Exclusion Criteria:

Stroke Participants:

Stroke onset more than 3 months prior to study entry.

Acutely medically unwell as per medical team

Patient is unable to follow verbal commands or has global aphasia. Interpreters may be used to accommodate stroke survivors' communication needs.

Severe illness with a life expectancy of less than 3 months (e.g., cancer, endocarditis, metastasis with an occult primary malignancy).

Uncontrolled hypertension as assessed by the treating physician.

Unstable angina or recent myocardial infarction.

Any history of epilepsy or seizures, except for febrile seizures of childhood.

Current participation in another clinical trial involving rehabilitation (e.g., recreational therapy, occupational therapy, physiotherapy) or an investigational drug that might interfere with study results.

Patient is unwilling or unable to comply with the protocol or cannot/will not cooperate fully with the investigator or study personnel.

Any physical health condition, mental health condition, or other medical condition or diagnosis that might confound the interpretation of results or put the patient at risk (e.g., amputation of one extremity).

History of vertigo.

Active delirium/significant levels of confusion

Cervical artery dissection.

Patients with implanted devices such as pacemakers, defibrillators, and cochlear implants.

Individual currently being managed under the Mental Capacity Act

Staff participants:

Uncontrolled hypertension as assessed by the treating physician.

Unstable angina or recent myocardial infarction

Any history of epilepsy, seizures, except for febrile seizures of childhood.

Current participation in another clinical trial involving rehabilitation (e.g., recreational therapy, occupational therapy, physiotherapy) or an investigational drug that might interfere with study results.

Any physical health condition, mental health condition, or other medical condition or diagnosis that might confound the interpretation of results or put the patient at risk (e.g., amputation of one extremity).

History of vertigo.

Cervical artery dissection.

Staff members with implanted devices such as pacemakers, defibrillators, and cochlear implants.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
System Usability Scale | Day 1 & Day 30
  Scale assess the usability of the resynk VR system for both arms higher score mean higher usability
Safety and Acceptability Questionnaire | Day 1 & Day 30
  A custom Questionnaire to evaluate the safety and acceptability of Resynk VR in both arms

SECONDARY OUTCOMES:
Upper limb function (Fugl-Meyer Assessment) | Day 1 & Day 30
  The standardised Fugl meyer upper limb assessment to assess upper limb function stroke survivor arm only
Quality of life (EQ-5D-5L) | Day 1 & Day 30 & Day 60
  Assess the quality of life of the patient before and after intervention stroke survivor arm only
self-efficacy (General Self-Efficacy Scale) | Day 1 & Day 30
  self-efficacy is a person's perception of their ability to perform tasks stroke survivor arm only
rehabilitation intensity (resynk repetition count vs average conventional therapy based on literature) | Day 1 & Day 30
  Compare resynk rehab intensity vs conventional to show service improvement or not, stroke survivor arm only

CONTACTS AND LOCATIONS:
Overall Officials: Emma Dunn, Bsc, Principal Investigator — Belfast Health and Social Care Trust
Locations (1):
- Royal Victoria Hospital, Belfast, Down, United Kingdom

IPD SHARING:
Plan to Share IPD: No